CLINICAL TRIAL: NCT05357235
Title: The Clinical Outcome of Inactive HBsAg Carrier Patients With Low HBV DNA Levels and Normal ALT by Antiviral Therapy
Brief Title: The Study on Optimal Treatment and Clinical Outcome of Chronic Hepatitis B Patients With Inactive Hypoviremia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Collaborators: Beijing 302 Hospital/5th Medical Center of Chinese PLA General Hospital (Unknown); Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of the second Department of liver diseases, Beijing Ditan Hospital
Other Study IDs: CFH2022-1-2172-2
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B infection; Inactive HBsAg Carrier; Clinical Outcome; Nucleoside analogues
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment intervention group: NA (TDF or TAF) combined with PEG-IFN was used. PEG-IFN was injected subcutaneously once a week and a personalized course of 24 weeks was used.
  Interventions: Drug: PEG-IFN
- Non therapeutic intervention observation group: patients do not receive treatment and are observed and followed up regularly.

INTERVENTIONS:
Drug: PEG-IFN — PEG-IFN 180 or 135 micrograms, subcutaneously injected once a week, with a personalized treatment course of 24 weeks
  Groups: Treatment intervention group

SUMMARY:
Chronic hepatitis B seriously endangers the health of our people, especially the occurrence of HCC, which brings huge economic burden and life threat to our people. 84% - 92% of HCC in China is related to chronic HBV infection. How to further reduce the risk of liver cancer is an urgent problem to be solved in clinical research and an important direction. Although NAs treatment can make patients achieve the negative transformation of virus, it can not effectively reduce the level of virus antigen, and it also lacks the ability to improve the immune clearance of virus. As a result, the incidence of liver cancer in patients with long-term NA treatment is still 4.5% - 10.5%, and the incidence of HCC in patients with hypoviremia in Na treatment is higher. In current clinical practice, nearly 1 / 3 of patients treated with NAs can not reach the detection line of highly sensitive reagent. It is an important measure to make the patients with hypoviremia and inactive low virus replication treated by NAs below the detection line of highly sensitive reagent and further reduce the risk of HCC. However, it is still not enough to minimize the risk of HCC to achieve a complete viral response only through NA treatment. The long-term follow-up showed that the incidence of HBsAg disappeared by only 2.0% - 0.0% regardless of the long-term treatment of HBsAg. Therefore, the most important measure to minimize the occurrence of HCC is to optimize the treatment of NA treated patients with low virus replication and inactive patients with low virus replication to achieve complete virus response and clinical cure. The purpose of this study is to explore the optimal treatment scheme for chronic hepatitis B NA treated patients with hypoviremia and natural low virus replication patients to significantly reduce the risk of HCC.

DETAILED DESCRIPTION:
Chronic hepatitis B seriously endangers the health of our people, especially the occurrence of liver cancer, which brings huge economic burden and life threat to our people. 84% - 92% of hepatocellular carcinoma (HCC) in China is related to chronic HBV infection. How to further reduce the risk of liver cancer is an urgent problem to be solved in clinical research and an important direction. Although NAs treatment can make patients achieve the negative transformation of virus, it can not effectively reduce the level of virus antigen, and it also lacks the ability to improve the immune clearance of virus. As a result, the incidence of liver cancer in patients with long-term NA treatment is still 4.5% - 10.5%, and the incidence of HCC in patients with hypoviremia in Na treatment is higher. In current clinical practice, nearly 1 / 3 of patients treated with NAs can not reach the detection line of highly sensitive reagent. It is an important measure to make the patients with hypoviremia and inactive low virus replication treated by NAs below the detection line of highly sensitive reagent and further reduce the risk of HCC. However, it is still not enough to minimize the risk of HCC to achieve a complete viral response only through NA treatment. The long-term follow-up showed that the incidence of HBsAg disappeared by only 2.0% - 0.0% regardless of the long-term treatment of HBsAg. Therefore, the most important measure to minimize the occurrence of HCC is to optimize the treatment of NA treated patients with low virus replication and inactive patients with low virus replication to achieve complete virus response and clinical cure. The purpose of this study is to explore the optimal treatment scheme for chronic hepatitis B Na treated patients with hypoviremia and natural low virus replication patients to significantly reduce the risk of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 16 to 60;
* The positive time of HBsAg was 6 months,
* 48 weeks of treatment with ETV, TDF or TAF, including HBeAg positive and negative patients;
* High sensitive reagent was used to confirm that the low level of serum HBV DNA was 20 IU / ml-2000 IU / ml.
* Good compliance and sign informed consent.

Exclusion Criteria:

1. Patients with decompensated liver cirrhosis or previous decompensated liver cirrhosis;
2. Those who have used interferon within 6 months;
3. at the same time, it is associated with other virus infections, such as hepatitis A virus, hepatitis C virus, hepatitis D virus, hepatitis E virus, AIDS virus, etc;
4. in addition to hepatitis B, there are other serious physical and mental diseases, including uncontrolled primary kidney, heart, lung, vascular, neurological, digestive, severe metabolic diseases (such as uncontrolled hyperthyroidism, serious complications of diabetes and adrenal diseases), immune deficiency diseases, and severe infections;
5. Active or suspected malignant tumor or history of malignant tumor;
6. 6 months before enrollment or currently receiving corticosteroids, immunosuppressants and chemotherapeutic drugs;
7. Complicated with alcoholic liver disease, autoimmune liver disease and other liver diseases;
8. HBV resistant patients;
9. Other situations that the researcher believes are not suitable for inclusion.

PegIFN α Treatment contraindications:

1. Prohibited for known pairs α- Patients who are allergic to interferon, E. coli products, polyethylene glycol or any component of this product;
2. It is forbidden to be used in patients with autoimmune hepatitis;
3. Pregnant and lactating women;
4. Central nervous system diseases, mental diseases, uncontrolled epilepsy, non withdrawal of alcohol / drug abuse, decompensated liver cirrhosis, symptomatic heart disease, uncontrolled autoimmune diseases and severe thyroid function diseases;
5. Absolute neutrophil count before treatment ≤ 1.0 × 109 / L, platelet ≤ 80 × 109/L。

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Chronic Hepatitis B patients With Inactive Hypoviremia
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of HCC during the project study | 48 weeks
  Once the hepatitis attack (HBV DNA > 2000 IU / ml, ALT >40 U / L) is reached during the observation of inactive low virus replication HBsAg carriers, the researchers will communicate with the patients and take antiviral treatment, and continue to follow-up observation. All enrolled patients were included in the continuous follow-up cohort during the study period and after the end of the project.

SECONDARY OUTCOMES:
The negative conversion rate of HBV DNA after 48 weeks of treatment was optimized (below the detection line of highly sensitive detection reagent) | 48 weeks
  Once the hepatitis attack (HBV DNA > 2000 IU / ml, ALT >40 U / L) is reached during the observation of inactive low virus replication HBsAg carriers, the researchers will communicate with the patients and take antiviral treatment, and continue to follow-up observation. All enrolled patients were included in the continuous follow-up cohort during the study period and after the end of the project.
The incidence of HBsAg disappearance during the study period; | 48 weeks
  Once the hepatitis attack (HBV DNA >2000 IU / ml, ALT > 40 U / L) is reached during the observation of inactive low virus replication HBsAg carriers, the researchers will communicate with the patients and take antiviral treatment, and continue to follow-up observation. All enrolled patients were included in the continuous follow-up cohort during the study period and after the end of the project.
HBeAg seroconversion rate in HBeAg positive patients; | 48 weeks
  Once the hepatitis attack (HBV DNA > 2000 IU / ml, ALT> 40 U / L) is reached during the observation of inactive low virus replication HBsAg carriers, the researchers will communicate with the patients and take antiviral treatment, and continue to follow-up observation. All enrolled patients were included in the continuous follow-up cohort during the study period and after the end of the project.
Incidence of chronic hepatitis B during the study period | 48 weeks
  Once the hepatitis attack (HBV DNA > 2000 IU / ml, ALT >40 U / L) is reached during the observation of inactive low virus replication HBsAg carriers, the researchers will communicate with the patients and take antiviral treatment, and continue to follow-up observation. All enrolled patients were included in the continuous follow-up cohort during the study period and after the end of the project.
To study the incidence of complications such as cirrhotic ascites and upper gastrointestinal bleeding during long-term follow-up. | 48 weeks
  Once the hepatitis attack (HBV DNA > 2000 IU / ml, ALT > 40 U / L) is reached during the observation of inactive low virus replication HBsAg carriers, the researchers will communicate with the patients and take antiviral treatment, and continue to follow-up observation. All enrolled patients were included in the continuous follow-up cohort during the study period and after the end of the project.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology Division 2, Beijing Ditan Hospital, Beijing, Beijing Municipality, China